CLINICAL TRIAL: NCT00312936
Title: A Mindfulness Based Approach to HIV Treatment Side Effects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: R21AT003102-01 (NIH); R21AT003102-01 (NIH)
Record Dates: First submitted 2006-04-07; First posted 2006-04-11 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: HIV Infections
Keywords: Medication adherence; Medication compliance; Quality of Life; Stress reduction; mindfulness based stress reduction; HIV/AIDS; treatment experienced
MeSH Terms: conditions — HIV Infections; Medication Adherence; Acquired Immunodeficiency Syndrome | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wait List (No Intervention)
- MBSR (Experimental): 8 week mindfulness based stress reduction
  Interventions: Behavioral: Mindfulness-based Stress Reduction (MBSR)

INTERVENTIONS:
Behavioral: Mindfulness-based Stress Reduction (MBSR) — 8 week program
  Arms: MBSR

SUMMARY:
We are exploring the effect that an 8 week stress reduction program based in mindfulness practices will have on the experience of medication side effects reported by HIV-infected men and women taking antiretroviral therapy.

DETAILED DESCRIPTION:
As HIV treatments continue to advance, people living with HIV will inevitably be confronted with negative physical and emotional side effects. Side effects from antiretroviral therapy (ART) for HIV impact quality of life (QOL) and adherence to care, and they influence decisions about health care. With mortality rates from HIV dramatically reduced in the US, side effects emerge as one of the most critical factors in the HIV epidemic. Eliminating or reducing the negative impact of side effects may improve QOL, reduce missed days from work, and maximize benefit from treatment for people living with HIV. We propose a randomized controlled trial (RCT) to provide preliminary evidence of the efficacy of a Mindfulness-Based Stress Reduction (MBSR) intervention to remediate side effects and side effect-related distress. Decreases in medical and psychological symptoms have been observed following MBSR in a wide range of illness contexts, but the approach has not been applied to HIV treatment side effects. Our team brings together expertise in HIV treatment side effects research, MBSR research with HIV+ populations, and HIV clinical medicine. The proposed study maximizes resources from our funded research programs within one of the leading AIDS research institutions in the world. Relevant research entities supporting this proposal include the Center for AIDS Prevention Studies (CAPS), the Osher Center for Integrative Medicine (OCIM), the UCSF Center for AIDS Research (CFAR) and the UCSF AIDS Research Institute (ARI). We propose a randomized clinical trial of an 8-week program of MBSR with 100 HIV+ men and women on ART, as compared with a wait list control (n=50/group). Primary outcome will be side effect distress and frequency, and secondary outcomes will be QOL and medication adherence. The findings from this study, in conjunction with our ongoing research studies, will provide foundation and guidance, including effect size data, for larger studies of MBSR for HIV disease.

ELIGIBILITY:
Inclusion Criteria:

1. HIV+ serostatus, evidenced by letter from provider, or official HIV test results.
2. Currently (prior 30 days) on an acknowledged ART regimen.
3. Reporting a level of side effect-related bother for the previous 30 days at or above eight (corresponding to the 40th% in another sample) on the side effect and symptom distress scale used in other studies.1, 89
4. Ability to provide informed consent to be a research participant.
5. English speaking.

Exclusion Criteria:

1. Current enrollment in a behavioral coping or HIV adherence intervention research study or MBSR program. A list of such studies/programs is kept and updated throughout the study.
2. Severe cognitive impairment as assessed by trained interviewer and confirmed by PI;
3. Active psychosis as assessed by trained interviewer and confirmed by PI;
4. Indication of active substance abuse that would interfere with capacity to participate in MBSR.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2006-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Patient reported number and severity of ART side effects | 6 months

SECONDARY OUTCOMES:
Health related quality of life | 6 months
ART adherence | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mallory O Johnson, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- See also: Related Info — http://www.caps.ucsf.edu